CLINICAL TRIAL: NCT02776111
Title: The Use of Microfluidics and Transcriptomics to Implement Precision Medicine in Post Solid Organ Transplant Patients
Brief Title: Microfluidics and Transcriptomics in Post Solid Organ Transplant Patients
Status: Terminated | Type: Observational
Why Stopped: Funding
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201600231
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Immunosuppression
Keywords: Kidney Transplant
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 400 microliters of blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: Participants in this group will have a one time blood sample taken.
  Interventions: Other: Blood Sample
- Kidney Transplant Group: Participants in this group have had a kidney transplant and blood samples will be obtained as described in study plan

INTERVENTIONS:
Other: Blood Sample — A one time blood sample will be provided.
  Groups: Healthy Controls

SUMMARY:
The field of genomics is an exciting new field being applied in medicine. Its use in treating some cancers, sepsis and burn patients has been very promising. As knowledge of genomics and application of microarrays expands, researchers are developing more intelligent ways to provide individualized care for patients. The plan of this research study is to apply the use of genomics as a tool for transplant in several capacities.

This research study is designed to develop methods of isolating relevant cell types via microarray plates, then extracting mRNA samples of those cell types and capturing their genetic profile. This will be done with the blood of up to ten healthy donors. Once this ability has been demonstrated, the next step will be to use these testing in several capacities in transplant patients. The research study plan involves following the genetic profile of 26 kidney transplant patients. One group will be followed prospectively starting at baseline, and then at various set time points. A second group will be sampled with the occurrence of clinical events. These events include viral, bacterial, and fungal infection, WBC < 2.5 or biopsy proven rejection episodes or normal graft function. Thus, the intention of the study is to demonstrate how immunosuppression alters the expression of this genetic expression of these T cells. In doing so, the study will provide a better understanding of the specific and true immunosuppressed state for any given patient.

DETAILED DESCRIPTION:
The two specific aims of the research study are as follows: 1) Proof of concept with two parts. Firstly, the study plan is to prove that T cells that are very commonly involved in the immune response: CD2, CD3, CD4, and CD8 populations can be captured. These cells will be captured, lysed and their mRNA genomics will be mapped. The second part of the proof of concept will involve exposing the CD2, CD3, CD4 and CD8 populations ex vivo to various serum concentrations of tacrolimus - the main cornerstone immunosuppressive medication in solid organ transplant. Exposure of the three cell types to the various tacrolimus concentrations will demonstrate that there is testing that can detect mRNA transcripts corresponding to under, optimal and over immunosuppressed states. The quantify IL2 production of the three cell types under the various immunosuppressive conditions will then be measured. With these 2 parts of the first specific aim of the study, a technique that can readily and easily isolate the cell populations of interest from the transplant patients and can capture how these cell populations respond to immunosuppression at various concentrations will have been demonstrated. 2) The second specific aim of the research study is running this genomic profiling on kidney transplant recipients. For this portion of the study, there will be two cohorts. A cohort identified as the "prospective" group and a cohort labeled as the "event" group. For the prospective cohort, blood will be obtained from the patients at specific time points. Specifically, blood samples will be obtained in the pre-transplant setting when the patients present to the hospital for their transplant, then at post-kidney transplant day 0, 1, 2, 3 and 7 (+/- 1 day) and at day 14, 21, and 28 (+/-3 days). Blood samples will be obtained again at months 2, 3, 6, 9, and 12 (+/- 1 week ). For the second group, blood samples will be obtained at the time of "events", such as rejection, infection, etc., and apply the same series of tests to their blood. For this group, blood draws will be done at time 0(+/-1 day), at then at one week (+/-2 days), and at one, two and three months (+/-1 week) post time 0. There will be five blood samples collected per patient. For all patients, there will be a comparison of the standard collected clinical information on the patient - graft function, rejection, infection, immunosuppression levels - to the results of our transcriptomics. The culmination of the project will involve revealing how genomics of the specific types of T cells can more precisely reflect a patient's true immunosuppressed state by corresponding to high, optimal and low immunosuppressive clinical phenotypes, and thus allow transplant clinicians to more intelligently and accurately administer immunosuppressive medications.

This study will involve obtaining blood samples on the kidney transplant patients at the time in which they would otherwise have blood collected for standard clinical care. Consent will be obtained for the testing on their blood, but the patients will not suffer any additional pain or inconvenience of the testing. In coordination with the equipment and supplies currently being used by the trauma and critical care department's research, the investigators will organize the collection and running of the labs in a time efficient and minimally expensive way

ELIGIBILITY:
Inclusion Criteria:

Healthy Controls

* consent for blood draw

Kidney Transplant Group

* actively listed with the University of Florida Kidney Transplant Program (which has its own standards for active listing including not being pregnant),
* consent for blood draw

Exclusion criteria:

Healthy Control

* pregnancy,
* any known organ failure

Kidney Transplant Group

* none, exclusive to what is listed in inclusion criteria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Controls and Kidney Transplant Patients
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-26 (Actual)

PRIMARY OUTCOMES:
Genomics of the T-cells will be compared to the immunosuppressed state of kidney transplant patient. | 12 months
  Standard collected clinical information of patients will identify over, optimal and under immunosuppressive states (IS) in kidney transplant (txp) recipients. In txp care, the definition of IS is defined by the clinical picture of the patient. Patients who have infections are over immunosuppressed, patients who have rejection are under immunosuppressed. Patients with neither and good graft function with normal Cr & good urine output have optimal IS. The investigators hope to identify a genomic pattern of the mRNA of T cells that correlates with the clinical picture of over, under or optimal IS in a kidney txp patient. Blood will be collected at the time of the events & genomics will be run on the T cell mRNA from that blood of each type of patient. The specific T cell used (CD3, CD4 or CD8) will be determined by the proof of concept portion of the study. The investigators will update this portion of the study as this information is obtained after the proof of concept is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zarrinpar, MD, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoniades CG, Berry PA, Wendon JA, Vergani D. The importance of immune dysfunction in determining outcome in acute liver failure. J Hepatol. 2008 Nov;49(5):845-61. doi: 10.1016/j.jhep.2008.08.009. Epub 2008 Aug 21. PMID 18801592
- [Background] Benitez C, Lozano JJ, Fueyo AS. Gene expression profiling and transplantation tolerance in the clinic. Transplantation. 2009 Aug 15;88(3 Suppl):S50-3. doi: 10.1097/TP.0b013e3181af7d17. PMID 19667962
- [Background] Brouard S, Mansfield E, Braud C, Li L, Giral M, Hsieh SC, Baeten D, Zhang M, Ashton-Chess J, Braudeau C, Hsieh F, Dupont A, Pallier A, Moreau A, Louis S, Ruiz C, Salvatierra O, Soulillou JP, Sarwal M. Identification of a peripheral blood transcriptional biomarker panel associated with operational renal allograft tolerance. Proc Natl Acad Sci U S A. 2007 Sep 25;104(39):15448-53. doi: 10.1073/pnas.0705834104. Epub 2007 Sep 14. PMID 17873064
- [Background] Bruls T, Gyapay G, Petit JL, Artiguenave F, Vico V, Qin S, Tin-Wollam AM, Da Silva C, Muselet D, Mavel D, Pelletier E, Levy M, Fujiyama A, Matsuda F, Wilson R, Rowen L, Hood L, Weissenbach J, Saurin W, Heilig R. A physical map of human chromosome 14. Nature. 2001 Feb 15;409(6822):947-8. doi: 10.1038/35057177. PMID 11237018
- [Background] Cuenca AG, Gentile LF, Lopez MC, Ungaro R, Liu H, Xiao W, Seok J, Mindrinos MN, Ang D, Baslanti TO, Bihorac A, Efron PA, Cuschieri J, Warren HS, Tompkins RG, Maier RV, Baker HV, Moldawer LL; Inflammation and Host Response to Injury Collaborative Research Program. Development of a genomic metric that can be rapidly used to predict clinical outcome in severely injured trauma patients. Crit Care Med. 2013 May;41(5):1175-85. doi: 10.1097/CCM.0b013e318277131c. PMID 23388514
- [Background] de Jonge J, Kurian S, Shaked A, Reddy KR, Hancock W, Salomon DR, Olthoff KM. Unique early gene expression patterns in human adult-to-adult living donor liver grafts compared to deceased donor grafts. Am J Transplant. 2009 Apr;9(4):758-72. doi: 10.1111/j.1600-6143.2009.02557.x. PMID 19353763
- [Background] Ding R, Li B, Muthukumar T, Dadhania D, Medeiros M, Hartono C, Serur D, Seshan SV, Sharma VK, Kapur S, Suthanthiran M. CD103 mRNA levels in urinary cells predict acute rejection of renal allografts. Transplantation. 2003 Apr 27;75(8):1307-12. doi: 10.1097/01.TP.0000064210.92444.B5. PMID 12717221
- [Background] Feezor RJ, Oberholzer C, Baker HV, Novick D, Rubinstein M, Moldawer LL, Pribble J, Souza S, Dinarello CA, Ertel W, Oberholzer A. Molecular characterization of the acute inflammatory response to infections with gram-negative versus gram-positive bacteria. Infect Immun. 2003 Oct;71(10):5803-13. doi: 10.1128/IAI.71.10.5803-5813.2003. PMID 14500502
- [Background] Feezor RJ, Baker HV, Mindrinos M, Hayden D, Tannahill CL, Brownstein BH, Fay A, MacMillan S, Laramie J, Xiao W, Moldawer LL, Cobb JP, Laudanski K, Miller-Graziano CL, Maier RV, Schoenfeld D, Davis RW, Tompkins RG; Inflammation and Host Response to Injury, Large-Scale Collaborative Research Program. Whole blood and leukocyte RNA isolation for gene expression analyses. Physiol Genomics. 2004 Nov 17;19(3):247-54. doi: 10.1152/physiolgenomics.00020.2004. PMID 15548831
- [Background] Feezor RJ, Cheng A, Paddock HN, Baker HV, Moldawer LL. Functional genomics and gene expression profiling in sepsis: beyond class prediction. Clin Infect Dis. 2005 Nov 15;41 Suppl 7:S427-35. doi: 10.1086/431993. PMID 16237642
- [Background] Gentile LF, Cuenca AG, Efron PA, Ang D, Bihorac A, McKinley BA, Moldawer LL, Moore FA. Persistent inflammation and immunosuppression: a common syndrome and new horizon for surgical intensive care. J Trauma Acute Care Surg. 2012 Jun;72(6):1491-501. doi: 10.1097/TA.0b013e318256e000. PMID 22695412
- [Background] Hassan-Montero L, Bueno P, Olmedo C, Comino AM, Muffak-Granero K, Garcia-Alcalde F, Serradilla M, Villar JM, Garrote D, Blanco A, Ferron JA. Gene expression profiling in liver transplant recipients with alcoholic cirrhosis. Transplant Proc. 2008 Nov;40(9):2955-8. doi: 10.1016/j.transproceed.2008.08.085. PMID 19010158
- [Background] Heller RA, Schena M, Chai A, Shalon D, Bedilion T, Gilmore J, Woolley DE, Davis RW. Discovery and analysis of inflammatory disease-related genes using cDNA microarrays. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2150-5. doi: 10.1073/pnas.94.6.2150. PMID 9122163
- [Background] Huang Q, Liu D, Majewski P, Schulte LC, Korn JM, Young RA, Lander ES, Hacohen N. The plasticity of dendritic cell responses to pathogens and their components. Science. 2001 Oct 26;294(5543):870-5. doi: 10.1126/science.294.5543.870. PMID 11679675
- [Background] Huskey J, Gralla J, Wiseman AC. Single time point immune function assay (ImmuKnow) testing does not aid in the prediction of future opportunistic infections or acute rejection. Clin J Am Soc Nephrol. 2011 Feb;6(2):423-9. doi: 10.2215/CJN.04210510. Epub 2010 Nov 18. PMID 21088287
- [Background] Kim S, Park YM. Specific gene expression patterns in liver cirrhosis. Biochem Biophys Res Commun. 2005 Aug 26;334(2):681-8. doi: 10.1016/j.bbrc.2005.06.143. PMID 16009336
- [Background] Kotz KT, Xiao W, Miller-Graziano C, Qian WJ, Russom A, Warner EA, Moldawer LL, De A, Bankey PE, Petritis BO, Camp DG 2nd, Rosenbach AE, Goverman J, Fagan SP, Brownstein BH, Irimia D, Xu W, Wilhelmy J, Mindrinos MN, Smith RD, Davis RW, Tompkins RG, Toner M; Inflammation and the Host Response to Injury Collaborative Research Program. Clinical microfluidics for neutrophil genomics and proteomics. Nat Med. 2010 Sep;16(9):1042-7. doi: 10.1038/nm.2205. Epub 2010 Aug 29. PMID 20802500
- [Background] Kurian SM, Williams AN, Gelbart T, Campbell D, Mondala TS, Head SR, Horvath S, Gaber L, Thompson R, Whisenant T, Lin W, Langfelder P, Robison EH, Schaffer RL, Fisher JS, Friedewald J, Flechner SM, Chan LK, Wiseman AC, Shidban H, Mendez R, Heilman R, Abecassis MM, Marsh CL, Salomon DR. Molecular classifiers for acute kidney transplant rejection in peripheral blood by whole genome gene expression profiling. Am J Transplant. 2014 May;14(5):1164-72. doi: 10.1111/ajt.12671. Epub 2014 Apr 11. PMID 24725967
- [Background] Kurian SM, Fouraschen SM, Langfelder P, Horvath S, Shaked A, Salomon DR, Olthoff KM. Genomic profiles and predictors of early allograft dysfunction after human liver transplantation. Am J Transplant. 2015 Jun;15(6):1605-14. doi: 10.1111/ajt.13145. Epub 2015 Mar 31. PMID 25828101
- [Background] Larson AM. Palliative care for patients with end-stage liver disease. Curr Gastroenterol Rep. 2015 May;17(5):440. doi: 10.1007/s11894-015-0440-6. PMID 25855211
- [Background] Leventhal JR, Mathew JM, Salomon DR, Kurian SM, Friedewald JJ, Gallon L, Konieczna I, Tambur AR, Charette J, Levitsky J, Jie C, Kanwar YS, Abecassis MM, Miller J. Nonchimeric HLA-Identical Renal Transplant Tolerance: Regulatory Immunophenotypic/Genomic Biomarkers. Am J Transplant. 2016 Jan;16(1):221-34. doi: 10.1111/ajt.13416. Epub 2015 Jul 30. PMID 26227106
- [Background] Lin XC, Sui WG, Qi SW, Tang DE, Cong S, Zou GM, Zhang Y, Li H, Chen WB, Cheng ZQ, Dai Y. Quantitative proteomic profiling of renal tissue in human chronic rejection biopsy samples after renal transplantation. Transplant Proc. 2015 Mar;47(2):323-31. doi: 10.1016/j.transproceed.2014.10.010. PMID 25769567
- [Background] Llorent L, Richaud-Patin Y, Alcocer-Castillejos N, Ruiz-Soto R, Mercado MA, Orozco H, Gamboa-Dominguez A, Alcocer-Varela J. Cytokine gene expression in cirrhotic and non-cirrhotic human liver. J Hepatol. 1996 May;24(5):555-63. doi: 10.1016/s0168-8278(96)80140-1. PMID 8773910
- [Background] Luo Y, Shi B, Qian Y, Bai H, Chang J. Sequential monitoring of TIM-3 gene expression in peripheral blood for diagnostic and prognostic evaluation of acute rejection in renal graft recipients. Transplant Proc. 2011 Dec;43(10):3669-74. doi: 10.1016/j.transproceed.2011.08.106. PMID 22172823
- [Background] Martinez-Llordella M, Lozano JJ, Puig-Pey I, Orlando G, Tisone G, Lerut J, Benitez C, Pons JA, Parrilla P, Ramirez P, Bruguera M, Rimola A, Sanchez-Fueyo A. Using transcriptional profiling to develop a diagnostic test of operational tolerance in liver transplant recipients. J Clin Invest. 2008 Aug;118(8):2845-57. doi: 10.1172/JCI35342. PMID 18654667
- [Background] Mas VR, Fassnacht R, Archer KJ, Maluf D. Molecular mechanisms involved in the interaction effects of alcohol and hepatitis C virus in liver cirrhosis. Mol Med. 2010 Jul-Aug;16(7-8):287-97. doi: 10.2119/molmed.2009.00165. Epub 2010 Mar 26. PMID 20386865
- [Background] Mathias B, Lipori G, Moldawer LL, Efron PA. Integrating "big data" into surgical practice. Surgery. 2016 Feb;159(2):371-4. doi: 10.1016/j.surg.2015.08.043. Epub 2015 Oct 23. PMID 26603852
- [Background] Matignon M, Ding R, Dadhania DM, Mueller FB, Hartono C, Snopkowski C, Li C, Lee JR, Sjoberg D, Seshan SV, Sharma VK, Yang H, Nour B, Vickers AJ, Suthanthiran M, Muthukumar T. Urinary cell mRNA profiles and differential diagnosis of acute kidney graft dysfunction. J Am Soc Nephrol. 2014 Jul;25(7):1586-97. doi: 10.1681/ASN.2013080900. Epub 2014 Mar 7. PMID 24610929
- [Background] Menon MC, Keung KL, Murphy B, O'Connell PJ. The Use of Genomics and Pathway Analysis in Our Understanding and Prediction of Clinical Renal Transplant Injury. Transplantation. 2016 Jul;100(7):1405-14. doi: 10.1097/TP.0000000000000943. PMID 26447506
- [Background] Mira JC, Szpila BE, Nacionales DC, Lopez MC, Gentile LF, Mathias BJ, Vanzant EL, Ungaro R, Holden D, Rosenthal MD, Rincon J, Verdugo PT, Larson SD, Moore FA, Brakenridge SC, Mohr AM, Baker HV, Moldawer LL, Efron PA. Patterns of gene expression among murine models of hemorrhagic shock/trauma and sepsis. Physiol Genomics. 2016 Feb;48(2):135-44. doi: 10.1152/physiolgenomics.00072.2015. Epub 2015 Nov 17. PMID 26578697
- [Background] Modena BD, Kurian SM, Gaber LW, Waalen J, Su AI, Gelbart T, Mondala TS, Head SR, Papp S, Heilman R, Friedewald JJ, Flechner SM, Marsh CL, Sung RS, Shidban H, Chan L, Abecassis MM, Salomon DR. Gene Expression in Biopsies of Acute Rejection and Interstitial Fibrosis/Tubular Atrophy Reveals Highly Shared Mechanisms That Correlate With Worse Long-Term Outcomes. Am J Transplant. 2016 Jul;16(7):1982-98. doi: 10.1111/ajt.13728. Epub 2016 Mar 15. PMID 26990570
- [Background] Muffak-Granero K, Olmedo C, Garcia-Alcalde F, Comino A, Villegas T, Villar JM, Garrote D, Blanco A, Bueno P, Ferron JA. Gene network profiling before and after transplantation in alcoholic cirrhosis liver transplant recipients. Transplant Proc. 2012 Jul-Aug;44(6):1493-5. doi: 10.1016/j.transproceed.2012.05.017. PMID 22841193
- [Background] Nacionales DC, Szpila B, Ungaro R, Lopez MC, Zhang J, Gentile LF, Cuenca AL, Vanzant E, Mathias B, Jyot J, Westerveld D, Bihorac A, Joseph A, Mohr A, Duckworth LV, Moore FA, Baker HV, Leeuwenburgh C, Moldawer LL, Brakenridge S, Efron PA. A Detailed Characterization of the Dysfunctional Immunity and Abnormal Myelopoiesis Induced by Severe Shock and Trauma in the Aged. J Immunol. 2015 Sep 1;195(5):2396-407. doi: 10.4049/jimmunol.1500984. Epub 2015 Aug 5. PMID 26246141
- [Background] Nau GJ, Richmond JF, Schlesinger A, Jennings EG, Lander ES, Young RA. Human macrophage activation programs induced by bacterial pathogens. Proc Natl Acad Sci U S A. 2002 Feb 5;99(3):1503-8. doi: 10.1073/pnas.022649799. Epub 2002 Jan 22. PMID 11805289
- [Background] Oetting WS, Schladt DP, Guan W, Miller MB, Remmel RP, Dorr C, Sanghavi K, Mannon RB, Herrera B, Matas AJ, Salomon DR, Kwok PY, Keating BJ, Israni AK, Jacobson PA; DeKAF Investigators. Genomewide Association Study of Tacrolimus Concentrations in African American Kidney Transplant Recipients Identifies Multiple CYP3A5 Alleles. Am J Transplant. 2016 Feb;16(2):574-82. doi: 10.1111/ajt.13495. Epub 2015 Oct 20. PMID 26485092
- [Background] Pons JA, Revilla-Nuin B, Baroja-Mazo A, Ramirez P, Martinez-Alarcon L, Sanchez-Bueno F, Robles R, Rios A, Aparicio P, Parrilla P. FoxP3 in peripheral blood is associated with operational tolerance in liver transplant patients during immunosuppression withdrawal. Transplantation. 2008 Nov 27;86(10):1370-8. doi: 10.1097/TP.0b013e318188d3e6. PMID 19034005
- [Background] Reeve J, Halloran PF, Kaplan B. Common errors in the implementation and interpretation of microarray studies. Transplantation. 2015 Mar;99(3):470-5. doi: 10.1097/TP.0000000000000691. PMID 25695786
- [Background] Sigdel TK, Bestard O, Tran TQ, Hsieh SC, Roedder S, Damm I, Vincenti F, Sarwal MM. A Computational Gene Expression Score for Predicting Immune Injury in Renal Allografts. PLoS One. 2015 Sep 14;10(9):e0138133. doi: 10.1371/journal.pone.0138133. eCollection 2015. PMID 26367000
- [Background] Smalling RV, Delker DA, Zhang Y, Nieto N, McGuiness MS, Liu S, Friedman SL, Hagedorn CH, Wang L. Genome-wide transcriptome analysis identifies novel gene signatures implicated in human chronic liver disease. Am J Physiol Gastrointest Liver Physiol. 2013 Sep 1;305(5):G364-74. doi: 10.1152/ajpgi.00077.2013. Epub 2013 Jun 27. PMID 23812039
- [Background] Sood S, Testro AG. Immune monitoring post liver transplant. World J Transplant. 2014 Mar 24;4(1):30-9. doi: 10.5500/wjt.v4.i1.30. PMID 24669365
- [Background] Sui W, Dai Y, Huang Y, Lan H, Yan Q, Huang H. Microarray analysis of MicroRNA expression in acute rejection after renal transplantation. Transpl Immunol. 2008 Apr;19(1):81-5. doi: 10.1016/j.trim.2008.01.007. Epub 2008 Feb 5. PMID 18346642
- [Background] Sui W, Lin H, Peng W, Huang Y, Chen J, Zhang Y, Dai Y. Molecular dysfunctions in acute rejection after renal transplantation revealed by integrated analysis of transcription factor, microRNA and long noncoding RNA. Genomics. 2013 Oct;102(4):310-22. doi: 10.1016/j.ygeno.2013.05.002. Epub 2013 May 15. PMID 23684794
- [Background] Vanzant EL, Hilton RE, Lopez CM, Zhang J, Ungaro RF, Gentile LF, Szpila BE, Maier RV, Cuschieri J, Bihorac A, Leeuwenburgh C, Moore FA, Baker HV, Moldawer LL, Brakenridge SC, Efron PA; Inflammation and Host Response to Injury Investigators. Advanced age is associated with worsened outcomes and a unique genomic response in severely injured patients with hemorrhagic shock. Crit Care. 2015 Mar 4;19(1):77. doi: 10.1186/s13054-015-0788-x. PMID 25880307
- [Background] Vitalone MJ, Sigdel TK, Salomonis N, Sarwal RD, Hsieh SC, Sarwal MM. Transcriptional Perturbations in Graft Rejection. Transplantation. 2015 Sep;99(9):1882-93. doi: 10.1097/TP.0000000000000809. PMID 26154388
- [Background] Wasmuth HE, Kunz D, Yagmur E, Timmer-Stranghoner A, Vidacek D, Siewert E, Bach J, Geier A, Purucker EA, Gressner AM, Matern S, Lammert F. Patients with acute on chronic liver failure display "sepsis-like" immune paralysis. J Hepatol. 2005 Feb;42(2):195-201. doi: 10.1016/j.jhep.2004.10.019. PMID 15664244